CLINICAL TRIAL: NCT06226142
Title: The Ultrasound-guided Versus Bronchoscopy-guided vs Ultrasound-bronchoscopy-guided Percutaneous Dilational Tracheostomy Trial - Standardization or Customization?
Brief Title: The Ultrasound-guided vs Bronchoscopy-guided vs Ultrasound-bronchoscopy-guided Percutaneous Tracheostomy Trial
Acronym: BRONCUS-PDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Constantinescu Catalin, Assistant lecturer, PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UMF-USBR-2024-001
Record Dates: First submitted 2024-01-05; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Tracheostomy Complication; Tracheostomy Infection; Tracheostomy Hemorrhage

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomized in a 1:1:1 ratio to ultrasound or bronchoscopy or ultrasound-bronchoscopy percutaneous dilatational tracheostomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound guided percutaneous tracheostomy (Experimental): The PDT will be performed by the attending physician exclusively with the aid of the ultrasound.
  Interventions: Procedure: Percutaneous dilatational tracheostomy
- Bronchoscopy guided percutaneous tracheostomy (Active Comparator): The PDT will be performed by the attending physician exclusively with the aid of the bronchoscope.
  Interventions: Procedure: Percutaneous dilatational tracheostomy
- Ultrasound-bronchoscopy guided percutaneous tracheostomy (Active Comparator): The PDT will be performed by the attending physician with the aid of the ultrasound and bronchoscope.
  Interventions: Procedure: Percutaneous dilatational tracheostomy

INTERVENTIONS:
Procedure: Percutaneous dilatational tracheostomy — Percutaneous dilatational tracheostomy

SUMMARY:
This trial (BRONCUS) is a randomized one designed to evaluate the overall safety of ultrasound guided compared to bronchoscopy guided compared to ultrasound-bronchoscopy guided percutaneous tracheostomy, in order to find out if universal standardization is required or customized approach can be sufficient.

DETAILED DESCRIPTION:
Enrolled patients will be randomized in a 1:1:1 ratio to ultrasound or bronchoscopy or ultrasound-bronchoscopy arms, and then the procedure related complications and clinical outcomes will be evaluated and compared between the groups. The procedures will be performed according to standardized practices following hospital guidelines.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (over 18 years old), intubated, mechanically ventilated, and with an indication for a tracheostomy

Exclusion Criteria:

Patients with contraindications for PDT:

* short neck
* tracheal deviation
* difficult anatomy
* previous neck surgery
* cervical trauma or inability to perform neck extension
* preference for surgical tracheostomy by the patient assistant team
* patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-01-06 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
PDT feasibility/failure | During PDT - 15-25 minutes
  Conversion to a surgical tracheostomy in any case, associated use of bronchoscopy in the case of ultrasound-guided PDT, associated use of ultrasound in the case of bronchoscopy-guided PDT, or the occurrence of a major complication.

SECONDARY OUTCOMES:
Minor complication - hypotension | During PDT (an expected average of 15-30 minutes)
  a drop of MAP<65 mmHg for less than 5 minutes without the requirement of fluids or vasopressors
Procedure difficulty | During PDT (an expected average of 15-30 minutes)
  (1) easy, (2) somewhat difficult, (3) difficult, (4) very difficult, or (5) impossible
ICU mortality | During hospital LOS (an expected average of 4 weeks )
  We will measure ICU mortality at the discharge and 60 days after discharge.
Hospital mortality | During hospital LOS (an expected average of 4 weeks)
  We will measure hospital mortality at the discharge and 60 days after discharge.
Procedure duration | During PDT (an expected average of 15-30 minutes)
  We will measure the procedure duration from the point beginning of the procedure and the end of it.
Mechanical ventilation | During hospital LOS (an expected average of 4 weeks)
  Days of MV before and after PDT
Minor complication - hypoxemia | During PDT (an expected average of 15-30 minutes)
  A drop in peripheral oxygen saturation < 90% for more than 2 minutes as measured by pulse oxymeter during the procedure while the patient is of 100% FiO2
Minor complication - Accidental decannulation | During hospital LOS (an expected average of 4 weeks)
  Accidental decannulation
Minor complication - Tracheostomy stoma infection | During hospital LOS (an expected average of 4 weeks)
  Tracheostomy stoma infection
Minor complication - Localized minor bleeding | During PDT (an expected average of 15-30 minutes)
  Localized minor bleeding
Minor complication - Localized subcutaneous emphysema | During PDT (an expected average of 15-30 minutes)
  Localized subcutaneous emphysema
Lenght of ICU stay | (an expected average of 4 weeks)
  Lenght of ICU stay
Lenght of hospital stay | (an expected average of 4 weeks)
  Lenght of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Petrisor, Prof, Study Chair — Iuliu Hatieganu University of Medicine and Pharmacy
Locations (1):
- Emergency County Clinical Hospital, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No